CLINICAL TRIAL: NCT05730686
Title: FibroLamellar Carcinoma: an International Registry Study
Acronym: FLiCIR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 22HH8014
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Fibrolamellar Cancer of the Liver

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Archival Tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Registry of Therapy of patient's diagnosed with FibroLamellar — Registry of Therapy of patient's diagnosed with FibroLamellar

SUMMARY:
Fibrolamellar Hepatocellular Carcinoma (FLC) is a rare (0.05 per 100,000) subtype of primary liver cancer which predominantly affects younger patients, median age of diagnosis 22-23 years. In patients with advanced stage disease the prognosis is poor, and even with aggressive surgery the 5 year survival is less than 50%.

Due to the very low incidence of FLC clinical trials are limited, and as these patients are excluded from most clinical trials there is a lack of consensus on the optimal systemic therapy to employ in this population group.

There are a number of chemotherapy compounds that have been investigated although these are single-institutional case series and/or registry-based studies. The majority of published registry studies are based in the United States hence it is important to describe the patterns of treatment in Europe which has different regulatory approvals for access to therapeutics. Our aim is to run a European multisite registry study detailing the clinical course of >100 patients with FLC that have received systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmed diagnosis of FLC
* Written informed consent will be required for the prospective cohort
* Adults of >18 years of age

Exclusion Criteria:

* Any non- histologic confirmed diagnosis of FLC
* Participants with insufficient clinical/ follow up data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective patients will be recruited from clinic
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
To describe the natural history and clinical outcomes of patients with Fibrolamellar carcinoma of the liver | 2 years
  The following data will be outcomes of interest in this study: treatments received including compliance and tolerability, survival (overall and progress free survival), clinicopathological outcomes. Survival outcomes, response rates